CLINICAL TRIAL: NCT07186179
Title: Mobilization of CD34+ Peripheral Blood Stem Cells With Filgrastim (Granulocyte-colony Stimulating Factor) and Plerixafor From Patients With Diamond Blackfan Anemia Syndrome
Brief Title: Mobilization of CD34+ Peripheral Blood Stem Cells in Patients With Diamond Blackfan Anemia Syndrome (DBAS)
Status: Recruiting | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Alexandra Satty, Assistant Professor Hofstra University/ Attending Physician Cohen Children's Medical Center, Northwell Health
Other Study IDs: 24-0953-CCMC
Record Dates: First submitted 2025-09-08; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Diamond Blackfan Anemia
Keywords: Diamond Blackfan Anemia; Mobilization; CD34+; GCSF
MeSH Terms: conditions — Anemia, Diamond-Blackfan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Mobilization Regimen — This study will utilize a standard mobilization regimen that is used for peripheral blood stem cell mobilization in patients with a variety of underlying conditions.
  Upon study initiation, participants will undergo a peripheral blood draw and bone marrow aspiration and biopsy. They will then begin the following mobilization regimen:
  1. Granulocyte-colony stimulating factor (G-CSF; filgrastim) dosed at 10mcg/kg/day administered subcutaneously in the morning for 5-7 days
  2. Plerixafor dosed at 0.24mg/kg/day administered subcutaneously in the evening for 1-4 days
  Participants will undergo daily blood draws until criteria for study completion is achieved.

SUMMARY:
Gene therapy is a new possible treatment for the anemia of DBAS. Gene therapy will soon be available for patients with RPS19-mutated DBAS. This involves inserting the corrected RPS19 gene into the cells, leading to correction of the anemia. The application of gene therapy requires sufficient numbers of stem cells on which the correction can be performed. Stem cells must be mobilized (stimulated to move) from the bone marrow to the peripheral blood and then collected (also called 'harvested'). It is not known if patients with DBAS can mobilize enough stem cells into the peripheral blood to allow for the harvesting of sufficient numbers to permit genetic manipulation. It is important to demonstrate the ability to harvest an adequate number of stem cells before gene therapy can be tried in patients with DBAS. The purpose of this study is to determine if mobilization of stem cells from the bone marrow in patients with DBAS is enough to obtain the numbers of peripheral blood stem cells necessary for effective gene therapy. An actual harvest will not be done.

DETAILED DESCRIPTION:
Diamond Blackfan anemia syndrome (DBAS) is a rare, inherited bone marrow failure syndrome, characterized by severe anemia, birth defects and a predisposition to cancer. The majority of patients with DBAS have a mutation in a gene encoding either a small (S) or large (L) subunit-associated ribosomal protein (RP). DBAS typically presents with severe anemia within the first two months of life. Approximately 80% of patients are initially responsive to corticosteroids with an improvement of their anemia, whereas 20% will not respond and will require red blood cell transfusions. Of the 80% of patients that initially respond to corticosteroid treatment, only about half of them will sustain a therapeutic response at a tolerable dose and the remainder will have to resort to transfusions for life. Overall ~20% of the patients may ultimately be able to discontinue corticosteroid or transfusion therapy and enter a treatment-independent phase. The only curative therapy for the anemia associated with DBAS at this time is allogeneic hematopoietic stem cell transplantation, however, this is limited by the availability of matched donors as well as the potentially life-threatening complications associated with transplantation.

There is a critical need for novel therapeutic options for these patients. Of the 28 known DBAS genes, RPS19 mutations are noted in 25% of patients. Gene therapy represents a potential curative option for the anemia of DBAS. This therapy involves inserting the corrected vector (in this case containing the RPS19 gene) into hematopoietic stem cells (HSCs), leading to correction of the anemia in animal models and, potentially, in humans. The application of gene therapy requires sufficient numbers of HSCs on which the correction can be performed. It has not been determined if patients with DBAS can mobilize enough HSCs into the peripheral blood to allow for the harvesting of sufficient numbers to permit genetic manipulation. It is important to demonstrate the ability to harvest an adequate number of HSCs before gene therapy can be contemplated for this rare population.

Patients with DBAS are known to have a reduced number of cells in the bone marrow, especially as the patients age, which raises the concern that HSCs may not be able to be mobilized into the peripheral blood. The goal of this project is to determine the feasibility of peripheral blood HSC collection in patients with DBAS to obtain the numbers necessary for effective gene therapy. Participants in this study will undergo bone marrow aspiration and biopsy to assess the cellularity and CD34+ cell count of the bone marrow, then begin a standard stem cell mobilization protocol consisting of filgrastim (granulocyte-colony stimulating factor, G-CSF; a white blood cell stimulating factor) and plerixafor. Participants will then undergo bloodwork by venipuncture to quantify the stem cell count in the peripheral blood to determine if enough stem cells can be collected. There will NOT be an actual stem cell collection. The study will also assess factors that may be predictive of successful peripheral blood HSC mobilization, including peripheral blood stem cell count, initial bone marrow cell number, and initial bone marrow CD34 count. The target population for this study will include individuals with a known DBAS mutation who are red blood cell transfusion dependent. The study aims to recruit a total of 10 participants between the ages of 3 and 30 years. At least 4 participants will be recruited with an RPS19 mutation and at least 6 participants will be under 18 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Diamond Blackfan anemia syndrome as defined by the known criteria with a known gene mutation
2. Male or female patients of all ethnic background, greater than or equal to 3 years of age and weighing at least 10 kg, and less than or equal to 30 years of age
3. Enrolled in Diamond Blackfan Anemia Registry of North America (DBAR)
4. Chronically red blood cell transfusion dependent for at least 6 months
5. Performance scale (Lansky Play-performance Scale for Pediatric Functional Status for age <16 years; Karnofsky Performance Scale for age ≥16 years) ≥ 70
6. Must sign informed consent

Exclusion Criteria:

1. Receiving prednisone therapy for treatment of DBAS (this does not include patients receiving physiologic steroid replacement for adrenal insufficiency)
2. Known history of myelodysplasia or presence of a hematopoietic clone
3. Current malignancy or previous treatment for malignancy
4. Pregnancy or breast-feeding mother
5. Known history of severe iron overload as defined by a liver iron concentration (LIC) > 15 mg Fe/ g dry liver weight
6. Significant cytopenias, defined as:

   * Platelet count <100,000/mcL
   * Absolute neutrophil count <750/mCL
7. Any GCSF use in the 3 months prior to enrollment
8. Liver dysfunction: aspartate aminotransferase (AST), alanine aminotransferase (ALT), or direct bilirubin values >3 x the upper limit of normal (ULN)
9. Kidney dysfunction: baseline estimated glomerular filtration rate (GFR) <70 mL/min/1.73 m2

Ages: 3 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Diamond Blackfan Anemia Syndrome (DBAS) ages 3-30 with red blood cell transfusion dependence
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of collecting 5-30 CD34+ cells/µL in patients ages 3 to 30 years with Diamond Blackfan anemia syndrome | 2 weeks
  This study will analyze the number of participants that successfully achieve 5-30 CD34+ cells/µL peripheral blood during the study period.

SECONDARY OUTCOMES:
Time to successful mobilization of CD34+ cells/µL peripheral blood | 2 weeks
  For participants who achieve a peripheral blood CD34+ count of 5-30/µL, the time (in days) from the start of mobilization regimen to successful mobilization (the day at which peripheral blood CD34+ count = 5-30/µL) will be quantified
Correlation of bone marrow CD34+ count with the ability to mobilize an adequate number of CD34+ cells in the peripheral blood. | 2 weeks
Correlation of mobilization of 5-30 CD34+ cells/µL peripheral blood with subject's age | 2 weeks
Correlation of mobilization of 5-30 CD34+ cells/µL peripheral blood with bone marrow cellularity. | 2 weeks
Correlation of mobilization of 5-30 CD34+ cells/µL peripheral blood with DBAS genotype | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Satty, MD, Principal Investigator — Northwell Health
Locations (1):
- Cohen Children's Medical Center, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No